CLINICAL TRIAL: NCT06993649
Title: Evaluation of Ability to Have a Normal Birth Using Different Simulation Methods: A Randomized Controlled Trial
Brief Title: Evaluation of Ability to Have a Normal Birth and Simulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Döndü BATKIN ERTÜRK, Assistant professor, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: TOKAT04
Record Dates: First submitted 2025-04-04; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Educational Problems
Keywords: normal birth skills; midwifery; simulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental High Reality simulator (Experimental): The steps of the process including normal labor skills will be done by each student in the d1= High Reality simulator (full-size, computer-based, time-adjusted, mother's statements about pain, performed with a female robotic simulator, Noelle S575 Mother and Newborn simulator)will be done to each student in the group respectively.
  Interventions: Behavioral: Experimental High Reality Simulator
- Experimental Medium Reality Simulator (Experimental): The steps of the process including normal labor skills will be done by each student in the d2= Medium Reality simulator (full-size, fetal heart sounds can be listened to, time-adjusted with a simple hand monitor, birth process performed with an automatic birth system, SB32878U full-size birth model) will be done to each student in the group respectively.
  Interventions: Behavioral: Experimental Medium Reality Simulator
- Experimental Simulated Woman (Experimental): The process steps including normal labour skills will be shown on d3= simulated woman (manual delivery of the baby, Gaumard S500 Half-Length Birth Simulator on which the midwifery student will apply the labour scenario) will be done to each student in the group respectively.
  Interventions: Behavioral: Experimental Simulated Woman

INTERVENTIONS:
Behavioral: Experimental High Reality Simulator — The process steps including normal labour skills will be shown on d1= High Reality simulator (full-size, computer-based, time-setting, expressions of pain from the mother, performed with a female robotic simulator, Noelle S575 Mother and Newborn simulator), d2= Medium Reality simulator (full-size, fetal heart sounds can be listened, SB32878U full-length birth model, timed with a simple hand-held monitor, birth process is performed with an automatic birth system) and d3= simulated woman (manual delivery of the baby, Gaumard S500 Half-Length Birth Simulator on which the midwifery student will apply the labour scenario) will be done to each student in the group respectively.
  Arms: Experimental High Reality simulator
Behavioral: Experimental Medium Reality Simulator — The process steps including normal labour skills will be shown on d2= Medium Reality simulator (full-size, fetal heart sounds can be listened, SB32878U full-length birth model, timed with a simple hand-held monitor, birth process is performed with an automatic birth system) will be done to each student in the group respectively.
  Arms: Experimental Medium Reality Simulator
Behavioral: Experimental Simulated Woman — Then, the process steps including normal labour skills will be shown d3= simulated woman (manual delivery of the baby, Gaumard S500 Half-Length Birth Simulator on which the midwifery student will apply the scenario of labour by the midwifery student) will be done to each student in the group respectively.
  Arms: Experimental Simulated Woman

SUMMARY:
The research is planned to be conducted in a randomized controlled design in order to determine the "Evaluation of Normal Birth Skills with Different Simulation Methods" of midwifery students.

DETAILED DESCRIPTION:
The midwifery profession is a combination of knowledge and skills. In this process, it is very important for educators to understand students' learning processes, know how to transfer practical applications to the clinical environment, and use different educational techniques. The increase in the number of students in midwifery education in Türkiye, the reduction of student density in hospitals especially during the pandemic period, limited suitable clinical practice areas and the low number of educators, patient safety, ethical and legal sanctions, etc. make it necessary to integrate different teaching techniques into education. Depending on these processes, educators should follow innovative educational techniques and strengthen the skills of students before they go to the clinic. In order to achieve these desired goals in students, simulation education techniques have been frequently used recently.

In the literature, simulation is defined as "a method that reflects a clinical situation as close to reality as possible and makes it easier to understand and manage when encountered in clinical practice". It is emphasized that simulated patient education reinforces theoretical knowledge and practice by providing students with a realistic clinical experience before they go to the clinic, is effective in gaining critical thinking, decision-making and psychomotor skills, and increases individual learning. In midwifery practice education, simulation can often be used to transfer knowledge, teach simple/complex technical skills, communication, teamwork and clinical decision-making processes.

In addition, simulation training has benefits in midwifery practices such as; Increasing their self-confidence, Developing clinical decision-making skills, Gaining experience by learning from their mistakes without harming patients, Reducing their anxiety about the clinic, Increasing the quality of their work, Achieving the ability to apply complete care, technical skills, decision-making, evaluation, teamwork and management skills .

Simulation is mostly preferred in the teaching of practical interventions. The acquisition of the ability to perform normal births, which is the basis of these practices, is one of the most important outcomes of the midwifery program.

However, the difficulties encountered during clinical education cause midwifery students to graduate without performing a sufficient number of independent normal births.The most important reason for these difficulties is the inadequacy of the application areas to meet the increasing number of students and the inadequacy of the number of women performing normal births due to the increasing number of cesarean births. However, in our country, midwifery students must fulfill the requirement of performing 40 normal births in order to graduate according to the provisions of the "Regulation on the Determination of Minimum Education Conditions for Medical, Nursing, Midwifery, Dentistry, Veterinary, Pharmacy and Architecture Education Programs" numbered 26775 and dated 2 February 2008.

The primary people responsible for normal birth are midwives. Therefore, the quality of the training to be given during midwifery education regarding the application of normal birth is extremely important. Midwifery students need to be competent both practically and theoretically before encountering a real case during birth. At the same time, since normal birth practice is a very complex practice, it can cause serious stress in the student due to the risks it carries.The high stress level of the student can cause the student to not respond effectively to stress and to fail in the application. Again, at this point, it is thought that performing these applications on simulators many times in order to reduce the effects of stress on the application can improve the situation.

Providing training for vaginal birth and emergency obstetric cases with simulation method can contribute to the reduction of malpractices, increase in team cooperation and coordination, increase in clinical decision-making skills within the team, increase maternal satisfaction during birth and increase in vaginal birth rates. Many studies have found that training with simulation in healthcare professionals increases knowledge and skills on vaginal birth and obstetric emergencies, increases self-confidence and learning satisfaction, provides a safe learning environment and contributes to the development of correct decision-making skills.When the simulation studies on midwifery skill training are examined, it has been found that skill training with simulation improves the learning, skills, teamwork, communication, decision-making and critical thinking skills of students in pregnancy, birth and emergency situations.

The research was conducted in a quasi-experimental randomized controlled design. The research will be conducted in the skill laboratories of the Midwifery Department of the Faculty of Health Sciences at Tokat Gaziosmanpaşa University.

The study will be conducted in the Department of Midwifery, Faculty of Health Sciences, during the 2024-2025 academic year. The sample of the study will consist of all third-year students (102 people) who registered for the Normal Birth and Postpartum Period course in the midwifery department for the first time. It is reported in the literature that in experimental studies, a sample size of at least 30 people is required to conduct parametric tests. In this study, the number of students in the groups was determined as 34 considering that there may be losses.

Students will be divided into three groups as d1= High Reality simulator, d2= Medium Reality simulator group and d3= simulated women group.

A total of 102 students will be studied. Students who meet the criteria for inclusion in the study will be given a sequence number and then randomly divided into 3 groups using the online randomization program https://www.randomizer.org.

Data Collection Tools In collecting the data; Introductory Information Form, Academic Motivation Scale and Student Satisfaction in Learning and Self-Confidence Scale will be used.

Introductory Information Form; It was created by the researchers by scanning the literature .This form consists of a total of 8 questions including the socio-demographic characteristics of the students, the presence of a health worker in the family, normal birth application status and characteristics related to simulation training (age, high school graduation, monthly income status, the presence of a health worker in the family, the status of receiving simulation training, etc.).

Motivation and Learning Strategies Scale This scale consists of two sections: Motivation Scale and Learning Strategies Scale .The Motivation Scale section of Motivation and Learning Strategies Scale was used to determine the criterion validity of the developed scale.The Motivation Scale consist of the factors of intrinsic goal regulation (items 1, 16, 22 and 24), extrinsic goal regulation (items 7, 11, 13 and 30), task value (items 4, 10, 17, 23, 26 and 27), self-efficacy perception regarding learning and performance (items 5, 6, 12, 15, 20, 21, 29 and 31), control belief regarding learning (items 2, 9, 18 and 25) and test anxiety (items 3, 8, 14, 19 and 28) factors.Cronbach alpha coefficients of the factors ranged between 0.86 and 0.41, and corrected item-total score correlation coefficients ranged between 0.19 and 0.66. Individuals mark their level of agreement with each statement on the scale on a seven-point rating scale ranging from "Absolutely False for Me" "1" to "Absolutely True for Me" "7". There is no cut-off point or reverse-scored item in the score calculation of the scale. A high score from any factor of the scale indicates that the student has a high level of the characteristic related to the said factor .

Student Satisfaction and Self-Confidence in Learning Scale;The original scale was developed as 13 items, and the total number of items was reduced to 12 during the adaptation to Turkish. The scale is a 5-point Likert-type scale and consists of the subheadings "Satisfaction with Current Learning" and "Self-confidence in Learning".

The subheading of satisfaction with current learning consists of 5 items, the subheading of self-confidence in learning consists of 7 items, and there are no negative items. The Cronbach alpha value of the scale for "Satisfaction with Current Learning" is .85, for "Self-confidence in Learning" it is .77, and for the total scale it is .89. Scale scores are obtained by dividing the sum of the sub-dimensions by the number of items.As the total score obtained from the scale increases, student satisfaction and self-confidence in learning also increase.

Application of the Research

All students taking the Normal Birth and Postpartum Period Course will be provided with the necessary information regarding normal birth practice within the scope of the course curriculum by the responsible lecturer of the course conducting the research, using the traditional learning method within the scope of slide presentation and video presentation.

At the end of the theoretical course; TBF will be applied to all students. After the theoretical lecture, normal labour skills training will be done in laboratory practice.

All students will be shown the process steps including normal labour skills on the simulator respectively by the instructor explaining the theoretical part of normal labour.

Then, the process steps including normal labour skills will be shown on d1= High Reality simulator (full-size, computer-based, time-setting, expressions of pain from the mother, performed with a female robotic simulator, Noelle S575 Mother and Newborn simulator), d2= Medium Reality simulator (full-size, fetal heart sounds can be listened, SB32878U full-length birth model, timed with a simple hand-held monitor, birth process is performed with an automatic birth system) and d3= simulated woman (manual delivery of the baby, Gaumard S500 Half-Length Birth Simulator on which the midwifery student will apply the labour scenario) will be done to each student in the group respectively.

Each group will work in different laboratories. Students will be taken to the laboratory practice by the same researcher in turns, without seeing each other.After the laboratory applications are completed, all students will be administered Motivation and Learning Strategies Scale and Student Satisfaction and Self-Confidence in Learning Scale . After the theoretical and laboratory parts of the course are completed, students will go to clinical practice for 8 weeks. After the clinical application, all students will be administered Motivation and Learning Strategies Scale and Student Satisfaction and Self-Confidence in Learning Scale again.

Statistical Analysis In the evaluation of the research data, Chi-Square Test (Chi Square Test) "paired sample t test in dependent groups", "independent sample t test" and Anova test will be used for intergroup evaluations.Statistical comparisons will be made with Mann-Whitney U-test and Wilcoxon Test. Variance Analysis or Friedman Variance Analysis will be used in Repeated Measures.The significance level will be accepted as p<0.05."

ELIGIBILITY:
Inclusion Criteria:

1. To be enrolled in Normal Birth and Postnatal Period Course for the first time
2. Not having participated in labour before
3. To volunteer to participate in the study

Exclusion Criteria:

1. To be enrolled in the Normal Birth and Postnatal Period Course for the second time

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-01-04 (Actual); Study Completion 2025-02-04 (Actual)

PRIMARY OUTCOMES:
Motivation Scale | one hour- two months
  "1" not at all true for me, "7" very true for me
Student Satisfaction and Self-Confidence in Learning Scale | one hour- two months
  1. "strongly disagree"
  2. "disagree"
  3. "undecided"
  4. "agree"
  5. "strongly agree"

CONTACTS AND LOCATIONS:
Overall Officials: Zümrüt YILAR ERKEK, Assoc. Prof., Principal Investigator — Tokat Gaziosmanpaşa University
Locations (1):
- Tokat Gaziosmanpaşa Üniversitesi, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lathrop A, Winningham B, VandeVusse L. Simulation-based learning for midwives: background and pilot implementation. J Midwifery Womens Health. 2007 Sep-Oct;52(5):492-8. doi: 10.1016/j.jmwh.2007.03.018. PMID 17826713
- [Background] Uyar Hazar, H., & Gültekin, S. (2019). Ebelik Eğitiminde Simülasyon Kullanımı, Life Sciences (NWSALS), 14(3), 74-83. DOI: 10.12739/NWSA.2019.14.3.4B0027.
- [Background] Edeer, A. D., & Sarikaya, A. (2015). The use of simulation in nursing education and simulation types/Hemsirelik egitiminde simulasyon kullanimi ve simulasyon tipleri. Journal of Education and Research in Nursing, 12(2), 121-126
- [Background] Nehring, W.M., & Lashley, F.R. (2009). Nursing simulation: A review of the past 40 years. Simulation & Gaming, 40(4), 528-552. https://doi.org/10.1177/1046878109332282
- [Background] Şendir, M. (2013). Use of simulation in women's health nursing education. F.N. Hem. Derg. 2013; 21(3): 205-212.
- [Background] Durmaz, A., Elem, E., Unutkan, A., & Keskin, N. (2017). The effect of simulation on vaginal delivery skills and self-sufficiency levels. J Curr Res Health Secto, 7(2), 41-52.
- [Background] Morgan PJ, Pittini R, Regehr G, Marrs C, Haley MF. Evaluating teamwork in a simulated obstetric environment. Anesthesiology. 2007 May;106(5):907-15. doi: 10.1097/01.anes.0000265149.94190.04. PMID 17457121
- [Background] Gardner R, Raemer DB. Simulation in obstetrics and gynecology. Obstet Gynecol Clin North Am. 2008 Mar;35(1):97-127, ix. doi: 10.1016/j.ogc.2007.12.008. PMID 18319131
- [Background] Göriş S., Bilgi N., Korkut Bayındır S. Hemşirelik Eğitiminde Simülasyon Kullanımı. Düzce Üniversitesi Sağlık Bilimleri Enstitüsü Dergisi 2014; 4 (2): 25-29
- [Background] Kamu Mevzuat Sistemi. https://kms.kaysis.gov.tr/Home/Goster/104346 erişim tarihi: 06.02.2018
- [Background] Demirel, G., Evcili, F., Kaya, N., Doganer, A. (2020). The effect of episiotomy repair simulation on the anxiety and self-efficacy levels of midwifery students. Journal of Midwifery and Reproductive Health, 8(1), 2050-2057. DOI: 10.22038/jmrh.2019.42024.1479
- [Background] DeStephano CC, Chou B, Patel S, Slattery R, Hueppchen N. A randomized controlled trial of birth simulation for medical students. Am J Obstet Gynecol. 2015 Jul;213(1):91.e1-91.e7. doi: 10.1016/j.ajog.2015.03.024. Epub 2015 Mar 12. PMID 25772212
- [Background] Crofts JF, Bartlett C, Ellis D, Hunt LP, Fox R, Draycott TJ. Training for shoulder dystocia: a trial of simulation using low-fidelity and high-fidelity mannequins. Obstet Gynecol. 2006 Dec;108(6):1477-85. doi: 10.1097/01.AOG.0000246801.45977.c8. PMID 17138783
- [Background] Dayal AK, Fisher N, Magrane D, Goffman D, Bernstein PS, Katz NT. Simulation training improves medical students' learning experiences when performing real vaginal deliveries. Simul Healthc. 2009 Fall;4(3):155-9. doi: 10.1097/SIH.0b013e3181b3e4ab. PMID 19680082
- [Background] Mert Karadas M, Terzioglu F. The impact of the using high-fidelity simulation and standardized patients to management of postpartum hemorrhage in undergraduate nursing students: A randomized controlled study in Turkey. Health Care Women Int. 2019 May;40(5):597-612. doi: 10.1080/07399332.2019.1583229. Epub 2019 Apr 2. PMID 30938581
- [Background] Lewis R, Strachan A, Smith MM. Is high fidelity simulation the most effective method for the development of non-technical skills in nursing? A review of the current evidence. Open Nurs J. 2012;6:82-9. doi: 10.2174/1874434601206010082. Epub 2012 Jul 27. PMID 22893783
- [Background] Hughes, C., Anderson, G., Patterson, D., & O'Prey, M. (2014). Introducing an obstetric emergency training strategy into a simulated environment. British Journal of Midwifery, 22(3), 201-207
- [Background] Arias T, Tran A, Breaud J, Fournier JP, Bongain A, Delotte J. A prospective study into the benefits of simulation training in teaching obstetric vaginal examination. Int J Gynaecol Obstet. 2016 Jun;133(3):380-4. doi: 10.1016/j.ijgo.2015.08.028. Epub 2016 Feb 23. PMID 26971257
- [Background] Yılar Erkek, Z., & Öztürk Altınayak, S. (2024, September). Assessing the Efficacy of Medium- and High-Reality Simulators in Normal Labor Management: A Randomized Controlled Trial. Clinical Simulation in Nursing, 94, 101599. https://doi.org/10.1016/j.ecns.2024.101599
- [Background] Yılar Erkek, Z., & Öztürk Altınayak, S. (2021, Month). The Effect of Simulation Teaching Technique on the Improvement of Episiotomy Performance Skills and State Anxiety of Midwifery Students in Turkey: RCT. Clinical Simulation in Nursing , 54, 62-69. https://doi.org/10.1016/j.ecns.2021.01.014 .
- [Background] Erkek, Z. Y., Alparslan, Ö., & Altınayak, S. Ö. (2021). The effect of simulation-based training about emergencies and approaches to delivery given to emergency personel. Clinical and Experimental Health Sciences, 11(1), 96-104.
- [Background] Carolan-Olah M, Kruger G, Brown V, Lawton F, Mazzarino M, Vasilevski V. Communicating out loud: Midwifery students' experiences of a simulation exercise for neonatal resuscitation. Nurse Educ Pract. 2018 Mar;29:8-14. doi: 10.1016/j.nepr.2017.10.027. Epub 2017 Oct 23. PMID 29144999
- [Background] Maskalova E, Urbanova E, Baskova M, Kvaltinyova E. Experience of lecturers with simulation training in midwifery education in Slovakia. Midwifery. 2018 Apr;59:1-3. doi: 10.1016/j.midw.2018.01.001. Epub 2018 Jan 5. PMID 29331775
- [Background] Özdamar, K. (2003). SPSS Statistical Package for the Social Sciences ile Bioistatistik. Eskişehir, Kaan Publisher.
- [Background] Khadivzadeh T, Erfanian F. The effects of simulated patients and simulated gynecologic models on student anxiety in providing IUD services. Simul Healthc. 2012 Oct;7(5):282-7. doi: 10.1097/SIH.0b013e31826064b7. PMID 22864014
- [Background] Khalaila R. Simulation in nursing education: an evaluation of students' outcomes at their first clinical practice combined with simulations. Nurse Educ Today. 2014 Feb;34(2):252-8. doi: 10.1016/j.nedt.2013.08.015. Epub 2013 Sep 3. PMID 24060462
- [Background] Unver V, Basak T, Watts P, Gaioso V, Moss J, Tastan S, Iyigun E, Tosun N. The reliability and validity of three questionnaires: The Student Satisfaction and Self-Confidence in Learning Scale, Simulation Design Scale, and Educational Practices Questionnaire. Contemp Nurse. 2017 Feb;53(1):60-74. doi: 10.1080/10376178.2017.1282319. Epub 2017 Feb 10. PMID 28084900
- [Background] Büyüköztürk, Ş., Akgün, Ö. E., Kahveci, Ö., & Demirel, F. (2004). Güdülenme ve öğrenme stratejileri ölçeğinin Türkçe formunun geçerlik ve güvenirlik çalışması. Kuram ve Uygulamada Eğitim Bilimleri, 4(2), 207-239.
- [Background] Shaw-Battista J, Belew C, Anderson D, van Schaik S. Successes and Challenges of Interprofessional Physiologic Birth and Obstetric Emergency Simulations in a Nurse-Midwifery Education Program. J Midwifery Womens Health. 2015 Nov-Dec;60(6):735-43. doi: 10.1111/jmwh.12393. Epub 2015 Dec 1. PMID 26624963